CLINICAL TRIAL: NCT03667781
Title: Pilot Study to Determine the Feasibility and Patient Acceptance of Therapeutic Drug Monitoring to Improve Medication Adherence
Brief Title: Therapeutic Drug Monitoring of Cardiac Medications
Status: Terminated | Type: Observational
Why Stopped: funding has ended and Covid has prevented us to perform followup assessment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 032018-023
Record Dates: First submitted 2018-09-04; First posted 2018-09-12 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Coronary Artery Disease
MeSH Terms: conditions — Hypertension; Coronary Artery Disease | interventions — Drug Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients Interviewed: Patients in cardiology clinic with uncontrolled hypertension despite being on 2 medications
- Providers Interviewed: Providers in cardiology clinic
- Patients Blood Draw: Patients seen in interventional clinic for post PCI followup will have a venous blood draw which will be sent for therapeutic drug monitoring
  Interventions: Diagnostic Test: Therapeutic drug monitoring

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring — Blood assay to evaluate for the presence of medications that the patient is prescribed. This is not being used for therapeutic purposes. It has already been validated in prior papers.
  Groups: Patients Blood Draw

SUMMARY:
The investigators will interview patients and providers of patients who have hypertension and are seen in cardiology clinic about ways to discuss therapeutic drug monitoring with patients. The investigators will use these interviews to crease discussion tools to discuss therapeutic drug monitoring. The investigators will then draw one venous blood sample in a different group of patients who are seen in interventional clinic for 1 month followup after PCI. The investigators will assay this blood for therapeutic drug monitoring and will provide the results to their providers for discussion at their regularly scheduled followup cardiology visit. The investigators will have the patients and providers fill out a survey afterwards to determine how they viewed therapeutic drug monitoring.

DETAILED DESCRIPTION:
The investigators will begin by conducting interviews with patients who have uncontrolled hypertension, defined as SBP>130 or DBP>80 mmHg despite treatment with > 2 antihypertensive drugs, from the Primary Care internal Medicine (PCiM) clinic and the cardiology clinic in the Parkland Health and Hospital System (Parkland). after obtaining informed consent for participation, we will explain therapeutic drug monitoring (TDM) as one method for accurately assessing the amount of prescribed antihypertensive medication in a patient's system and how that can be helpful to their physicians to effectively treat them. in these interviews, the investigators will assess reasons why patients may be nonadherent, why they may be reluctant to acknowledge this to their provider, explore how TDM could contradict patient self-report about adherence, how this contradiction could affect the patient-provider relationship, and how TDM could be used in a way that is acceptable to patients that enhances both the patient-provider relationship and improves patient health outcomes. The investigators anticipate conducting 10 interviews, after completing the patient interviews, the investigators will use what we have learned to guide the cognitive interviews with the hypertension clinicians. Provider participants will be recruited among physicians and nurses working in the PCiM and cardiology clinics at Parkland. The investigators will explore their responses to patient concerns, explore concerns about discussing and using TDM, especially how they might communicate the results of TDM testing that contradict patient self-reported medication adherence. After completing both patient and provider interviews, the investigators will create a TDM intervention discussion tool for providers to use and pilot this tool with a small group of TDM intervention pilot participants. This is an outline of the steps but the investigators will submit the surveys and discussion tools to the IRB for evaluation once they are developed. This will be done by a separate modification after the initial approval of the study once we have conducted the initial interviews. This group of participants will not be the same as the ones who were interviewed earlier. The discussion tool will include guidance to providers about explaining TDM and how it's useful for measuring adherence as well as prompts for addressing concerns patients identified in our interviews with them. The investigators will conduct this pilot intervention with 20 patients recruited from the PCiM and cardiology clinics who are being seen for their first follow-up visit post hospitalization, usually one month after discharge. Patients will be consented to participate in this TDM intervention, which will include measuring blood pressure, obtaining blood specimens for TDM, and eliciting patient self-report about medication adherence. Patients will be given their test results when they return for their next visit, usually 1-2 months later. although the blood assays for drug levels are not certified by CLIA nor approved by the FDA, the investigators are not using drug level information to change dosing or titrate the medications the patient are taking. During this second visit, the provider will then review the patient's TDM results and use the TDM discussion tool to guide conversation about discrepancies and potential barriers to adherence. The investigators will assess patients' reactions to and satisfaction with the discussion about TDM and its implications, and measure their blood pressure. Participants' reactions will be assessed by a survey tool.

The investigators will also assess perspectives about the patient's response to TDM and the effectiveness of using the TDM intervention discussion tool for facilitating the conversation with the patient. There are commercial assays that are FDA approved for used already. although the investigators do not use those assays, the Vanderbilt assays have been validated and published (though not approved by FDA).

ELIGIBILITY:
Inclusion Criteria:

Subjects age ≥ 18 to 80 years with uncontrolled hypertension (average clinic blood pressure of at least 130/80 mmHg despite treatment with 2 or more antihypertensive drugs).

Exclusion Criteria:

1. Presence of hypertensive emergency BP > 180/110 mmHg plus one of the following features: acute coronary syndrome, acute stroke, hypertensive encephalopathy, aortic dissection, or acute kidney injury,
2. History of active substance abuse such as alcohol, cocaine, or narcotics
3. Uncontrolled psychiatric disorder such as schizophrenia or major depression
4. Pregnancy
5. Homeless
6. Stage V CKD or end stage renal disease (glomerular filtration rate < 15 ml/min/1.73 m2),
7. Self-report of nonadherence or unwillingness to follow medication regimen prescribed by the primary care physicians for any reasons,
8. Presence of white coat hypertension (defined as normal 24-h ambulatory systolic BP or home BP of < 130 and diastolic BP of < 80 mmHg and clinic systolic BP of at least 140 mmHg or diastolic BP of at least 90 mmHg according to the AHA guidelines)
9. Inability to read or write English, because participants may not be able to follow all study procedures or complete study questionnaires and surveys correctly which may lead to inaccurate data collection.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients and providers seen in cardiology clinic for interview component. Patients seen in interventional clinic for their post PCI followup for the blood draw component.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Followup visit at 1 month from the initial visit
  Assessed by survey

SECONDARY OUTCOMES:
Provider Satisfaction | Followup visit at 1 month from the initial visit
  Assessed by survey

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No